CLINICAL TRIAL: NCT06296342
Title: Effects of Message Framing on Policy Support for Front-of-package Nutrition Labeling Among Latino and Limited English Proficiency Populations.
Brief Title: Message Framing and Policy Support for Front-of-package Labeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0300c
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2024-08

CONDITIONS: Diet, Healthy
Keywords: front-of-package labeling; policy support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No framing) (No Intervention): Participants will view one message about the front-of-package labeling policy. The message will display the same introductory sentence as all experimental arms, but it will not include a framed message about the objective of the front-of-package labeling policy.
- Information framing (Experimental): Participants will view one message that frames the objective of the front-of-package labeling policy as providing nutritional information.
  Interventions: Behavioral: Exposure to information framing message
- Healthier choices framing (Experimental): Participants will view one message that frames the objective of the front-of-package labeling policy as encouraging consumers to make healthier choices.
  Interventions: Behavioral: Exposure to healthier choices framing message
- Industry framing (Experimental): Participants will view one message that frames the objective of the front-of-package labeling policy as encouraging the food industry to make healthier products.
  Interventions: Behavioral: Exposure to industry framing message

INTERVENTIONS:
Behavioral: Exposure to information framing message — The information framing message presents the objective of the front-of-package labeling policy as providing nutritional information.
  Arms: Information framing
Behavioral: Exposure to healthier choices framing message — The healthier choices framing message presents the objective of the front-of-package labeling policy as encouraging consumers to make healthier choices.
  Arms: Healthier choices framing
Behavioral: Exposure to industry framing message — The industry framing message presents the objective of the front-of-package labeling policy as encouraging the food industry to make healthier products.
  Arms: Industry framing

SUMMARY:
This study aims to assess whether different message framing about front-of-package labeling policies elicits more policy support than the control (no framing) among Latino and limited English proficiency populations. The study also seeks to identify which message framing elicits the most policy support.

DETAILED DESCRIPTION:
Participants will complete a between-subjects online randomized experiment. Participants will be randomized to 1 of 4 arms: 1) No framing (control), 2) Information framing, 3) Healthier choices framing, and 4) Industry framing. In each arm, participants will view 1 message developed for their randomly assigned arm and indicate their policy support.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as Latino or Hispanic
* Ages 18-55 years old
* Residing in the United States

Exclusion Criteria:

* Not identifying as Latino or Hispanic
* Less than 18 or greater than 55 years old
* Not residing in the United States

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4107 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Support for the front-of-package labeling policy, proportion | During exposure to intervention (i.e., message about policy), assessed during one-time online 10-minute survey.
  Policy support will be assessed with 1 item: "How much would you support or oppose this policy?" This item will be measured on a 4-point scale ranging from (1) "Strongly oppose this policy" to (4) "Strongly support this policy", where higher scores indicate higher support for the front-of-package labeling policy. The final outcome will be dichotomized so that 0=Oppose this policy and 1=Support this policy.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill's Gillings School of Global Public Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared prior to data collection. After data collection and analysis, a de-identified version of individual participant data and the analytic code will be shared through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol and SAP will be available by mid-March 2024 (prior to data collection). IPD and analytic code will become available after data collection and analysis.
Access Criteria: Open access.